CLINICAL TRIAL: NCT02812368
Title: Clonidine for Sleep Disturbances in Children With Autism Spectrum Disorder
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Failure to recruit
Sponsor: Ohio State University (Other)
Collaborators: Autism Treatment Network (Network); Autism Intervention Research Network on Physical Health (Unknown)
Responsible Party: Principal Investigator, Jill Hollway, Assistant Professor of Research in Psychiatry, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016H0181
Record Dates: First submitted 2016-06-14; First posted 2016-06-24 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-01

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clonidine (Experimental): Taken once a day at bedtime; with the dose titrated from 0.05mg to 0.20mg over the course of 6 weeks
  Interventions: Drug: Clonidine
- Placebo (for clonidine) (Placebo Comparator): Taken once a day at bedtime
  Interventions: Drug: Placebo (for clonidine)

INTERVENTIONS:
Drug: Clonidine
  Other Names: Catapres, Kapvay, Duraclon
  Arms: Clonidine
Drug: Placebo (for clonidine) — Placebo pill manufactured to mimic clonidine
  Arms: Placebo (for clonidine)

SUMMARY:
Sleep disturbance has been reported in 44-86% of children with autism spectrum disorder (ASD) and is the source of considerable stress for the affected individual and family. Sleep plays a role in development and learning processes; thus, the appropriate treatment of sleep disturbance is paramount to optimal outcomes. The empirical base for treatments to address sleep in ASD is sparse, despite wide use of pharmacologic agents such as clonidine (CLN) to target sleep disturbance. A randomized, controlled pilot investigation of CLN for sleep disturbance in children with ASD will allow investigators to evaluate the feasibility of conducting a much larger multisite trial to address the general lack of systematic data available to guide practitioners. Subjects will be 16 children, ages 6-14 years, inclusive, with sleep disturbance and ASD. This randomized double-blind, placebo-controlled (PBO), parallel groups study will test the efficacy of CLN following a brief sleep hygiene intervention. Outcome measures include: informant completed sleep questionnaires, daytime behavior questionnaires, and actigraphy. Biomarkers for medication response will include galvanic skin response and skin temperature. Side effects will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* outpatients between 6-14 years of age, inclusive, from underserved populations (i.e., Low SES, racial and ethnic minorities, rural populations);
* diagnosis of Autism Spectrum Disorder based on DSM-V criteria and the ATN assessment protocol;
* mental age ≥ 24 months as determined by the Stanford Binet-Fifth Edition (SB-5) or Mullen Scales of Early Learning (MSEL) (the child must be of a mental age to understand the BI/SH protocol);
* significant sleep disturbance as determined the CSHQ 33-item Total Score of ≥ 48 and one of the following for the past four weeks by parent interview;

  1. ≥ 30 minutes delayed sleep onset, ≥ 3 times per week
  2. Sleep association problems, ≥ 3 nights per week, child falls asleep in a location other than his/her bed and requires parental intervention to return to his/her bed
  3. Nighttime Awakenings, ≥ 3 times per week, and child disturbs parent or enters into the parents' bedroom.
  4. Early Morning Awakenings, before 5 am ≥ 3 times per week and the child disturbs family members
* CGI Severity rating of ≥ 4 (Moderate) by the independent evaluator for sleep onset and/or sleep maintenance disruption at BL 2;
* care provider who can reliably bring subject to clinic visits and provide trustworthy ratings;
* stable dose of psychotropic medications (for at least 4 weeks with no plans to change over the course of the study);
* anticonvulsant if used for mood lability and it is working well;
* stable dose of exogenous melatonin for at least 4 weeks with no plans to change over the course of the study, as long as Phase II eligibility criteria are met prior to enrollment;
* sleep hygiene education responders who have relapsed and meet the Phase II study eligibility criteria

Exclusion Criteria:

* DSM-V diagnosis of bipolar disorder;
* subjects who are either melatonin naïve or who have not had an adequate trial of exogenous melatonin (defined as 3-5 mg for ≥ 4 weeks);
* seizure disorder/epilepsy;
* significant physical illness (e.g., serious cardiovascular, liver or renal pathology);
* medications specifically given for insomnia;
* pregnancy or sexually-active females without birth control;
* taking supplements or other complementary medical treatments where dose cannot be held at current level for duration of study;
* weight less than 15 kg;
* use of medicines for physical ailments that might interact with CLN or TRZ, such as guanfacine (Tenex, Intuniv), and propranolol (Inderol) or extended release clonidine (Kapvay);
* allergy to CLN or TRZ;
* Sleep Disordered Breathing (SDB) as defined by a total score of ≥ 3 on the CSHQ SDB subscale and parent report;
* prior adequate trial of CLN for sleep disturbance defined as at least 0.2mg q hs for 1 week;
* prior adequate trial of TRZ for sleep disturbance defined as ≥ 50 mg/day for 1 week;
* hyperthyroidism

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change in Children's Sleep Habits Questionnaire (CSHQ) Total Score | Change from Baseline to 6 Weeks
  The primary outcome measure for this study is clinical improvement on the CSHQ (defined as a 30% or greater reduction in the Total Score of the 33 Sleep Items) at 6 weeks compared to baseline. The CSHQ is the most commonly used parent-rated scale to assess sleep disturbance in pediatric populations. It includes 33 items and is rated retrospectively over the previous week by parents to screen for the most common sleep problems. The CSHQ incorporates items related to eight key sleep domains. The eight subscales include: (1) bedtime resistance (2) sleep onset latency, (3) sleep duration, (4) anxiety around sleep, (5) night awakenings, (6) sleep disordered breathing, (7) parasomnias and (8) morning waking/daytime sleepiness. A Total Score of 41 or greater on the CSHQ 33 items has been reported to be an appropriate clinical cut-off for identifying sleep problems in children.

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio State University Nisonger Center, Columbus, Ohio, United States